CLINICAL TRIAL: NCT01793402
Title: Adequacy of Vitamin D Intake and Vitamin D Status in Early Preterm Infants
Brief Title: Vitamin D Status and the Adequacy of Vitamin D Intake in Early Preterm Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Dr. Henry Akinbi, Associate Professor, Children's Hospital Medical Center, Cincinnati
Other Study IDs: VitD_Preterm#1
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants born at or less than 32 weeks gestation

SUMMARY:
Vitamin D is an essential nutrient. Deficiency of vitamin D is widespread. The prevalence of vitamin D deficiency in early preterm infants is unknown. The American Academy of Pediatrics recommends a daily intake of 400 IU in order to achieve a serum concentration of 20 ng/ml of vitamin D. This recommendation presumes exposure to sunlight, the best source of vitamin D. This study assesses vitamin D status at birth and during hospital stay in infants delivered delivered at earlier than or at 32 weeks gestation. We also assess the adequacy of intake relative to the target set by the American Academy of Pediatrics for children.

DETAILED DESCRIPTION:
Vitamin D is important for bone health. Deficiency of vitamin D is widespread and is associated with a variety of diseases. Preterm infants are susceptible osteopenia of prematurity (OP). Vitamin D deficiency may contribute to OP. The American Academy of Pediatrics (AAP) recommends a daily intake of 400 IU in order to achieve a serum concentration of 20 ng/ml of vitamin D. This recommendation presumes exposure to sunlight, the best source of vitamin D. Whether this level of intake or target serum concentration are achieved in early preterm infants is unknown. We hypothesize that because early preterm infants are sequestered in the Newborn Intensive Care Units for an extended period of time, they will be deficient in vitamin D and that the current nutritional intake may not be adequate in meeting the AAP recommendation. We assessed the concentration of serum 25-hydroxyvitamin-D in parturient mothers and in their newborns if they were less than 32 week gestation. We monitored vitamin D intake during hospitalization in the Newborn Intensive Care Unit and serum 25-hydroxyvitamin-D at discharge.

ELIGIBILITY:
Inclusion Criteria:

* All neonates delivered at or less than 32 weeks gestation were eligible.

Exclusion Criteria:

* Infants with lethal congenital malformation
* Infants that were not expected to survive to discharge
* Infants delivered from multiple gestation

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants born at or less than 32 weeks postmenstrual age admitted to the Newborn Intensive Care Unit at University of Cincinnati Medical Center were eligible. Intake of vitamin D and serum 25-hydroxyvitamin-D concentrations were assessed during stay in the Newborn Intensive Care Unit.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin-D concentration at the time of birth and at discharge from the hospital. | 6 weeks
  This is a longitudinal study that assessed vitamin D status at birth in infants as well as in their mothers. Daily intake of vitamin D was analyzed. The serum concentration of 25-hydroxyvitamin-D at discharge was assessed. We correlated maternal vitamin D with infants' vitamin D concentrations at birth. We also correlated vitamin D concentration at birth with the concentration at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Henry T Akinbi, M.D., Study Director — Children's Hospital Medical Center, Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States